CLINICAL TRIAL: NCT00823823
Title: Randomized Trial of Bivalved and Circumferential Casting for Displaced Forearm Fractures in Children
Brief Title: Randomized Trial of Casting Techniques for Displaced Forearm Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Donald Bae, Associate Professor of Orthopaedic Surgery, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-09-0430
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Displaced Forearm Fractures
Keywords: Casting techniques; Bivalved cast; Circumferential cast; Displaced distal radius fracture; Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bivalved cast (Active Comparator): Patients with a displaced distal radius or mid-diaphyseal forearm fracture requiring closed reduction will be immobilized in a bivalved cast
  Interventions: Other: Bivalved cast
- Circumferential cast (Active Comparator): Patients with a displaced distal radius or mid-diaphyseal forearm fracture requiring closed reduction will be immobilized in a circumferential cast
  Interventions: Other: Circumferential cast

INTERVENTIONS:
Other: Bivalved cast — Circumferential cast will be applied following closed reduction and then bivalved using a cast saw
  Arms: Bivalved cast
Other: Circumferential cast — Circumferential cast will be applied following closed reduction
  Arms: Circumferential cast

SUMMARY:
It is recognized that fractures of the distal radius and forearm occur in approximately one in 100 children and adolescents every year. Though closed manipulation and cast immobilization of displaced injuries is the mainstay of treatment in the majority of cases, the optimal type of cast remains debatable. Though well-molded casts theoretically provide the best ability to maintain fracture alignment, risks of circumferential immobilization in acute injuries include neurovascular compromise. Splitting, or bivalving, casts may reduce these risks, but the effect on fracture stability is unknown. The proposed investigation seeks to address the simple question of whether circumferential or bivalved casts provide the best outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Displaced distal radius or mid-diaphyseal forearm fracture
* fracture requires closed reduction and cast immobilization
* Age 4-16 years
* Skeletally immature

Exclusion Criteria:

* Failed closed reduction
* Acute fracture > 1 week old
* Refracture injury
* Fracture requires surgical treatment
* Significant soft tissue swelling
* Associated neurovascular compromise
* Plastic deformation injuries

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Bae, MD, Principal Investigator — Childrens Hospital Boston
Locations (1):
- Childrens Hospital Boston, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bivalved Cast | Circumferential Cast
Started | 109 | 107
Completed | 101 | 101
Not Completed | 8 | 6
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bivalved Cast | Circumferential Cast | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 101 | 101 | 202
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (6) | 10 (6) | 10 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 67 | 68 | 135
Region of Enrollment [Number; unit: participants]
  United States | 101 | 101 | 202

OUTCOME MEASURES:

1. Primary Outcome: Loss of Radius Fracture Reduction
Description: The number of participants that experienced radiographic loss of reduction by four weeks post-randomization.
Time Frame: 4 weeks post-randomization
Population: All subjects who completed the four-week follow-up period with no protocol violations.
Measure: Number; unit: participants
Arm/Group | Bivalved Cast | Circumferential Cast
Number analyzed (Participants) | 101 | 101
participants
  Loss of reduction | 35 | 35
  No Loss of reduction | 66 | 66
Statistical Analysis 1: Comparison: Bivalved Cast vs Circumferential Cast; The frequency of loss of reduction during the study period was compared across casting groups using a two-sided chi-square test with alpha = 0.05; Test type: Superiority or Other; p = 1.00, Chi-squared

2. Secondary Outcome: Compartment Syndrome or Neurovascular Compromise, Saw Burns and/or Lacerations
Description: The number of participants that experienced compartment syndrome or neurovascular compromise, saw burn and/or laceration within four weeks post-randomization.
Time Frame: Up to 4 weeks post-randomization
Population: All subjects who completed the four-week follow-up period with no protocol violations.
Measure: Number; unit: participants
Arm/Group | Bivalved Cast | Circumferential Cast
Number analyzed (Participants) | 101 | 101
participants
  Compartment syndrome | 0 | 0
  Cast saw burn | 0 | 0
  Laceration | 0 | 0
  Infection | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 6 weeks (from time of ED visit to last clinical follow-up visit)
Arm/Group | Bivalved Cast | Circumferential Cast
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/107
Other Adverse Events (participants affected / at risk) | 1/109 | 0/107
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bivalved Cast (N=109) | Circumferential Cast (N=107)
Cast saw burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No